CLINICAL TRIAL: NCT06051760
Title: A Phase I Study to Explore the Safety and Efficacy of NV-001 in the Treatment of Advanced Solid Tumors
Brief Title: NV-001 in the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NING LI, Director of Department of Clinical Trial Center, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV-001
Record Dates: First submitted 2023-07-26; First posted 2023-09-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Malignant Neoplasm
Keywords: Advanced solid tumor; Tumor vaccine
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NV-001 (Experimental): The patients will be treated with vaccines generated based on their tumor tissues.Various doses will be tested according to the protocol.
  Interventions: Biological: NV-001

INTERVENTIONS:
Biological: NV-001 — NV-001 is a type of tumor vaccine generated by hybridization of the tumor cell membrane and adjuvant membrane to stimulate the immune reactions against cancer cells.

SUMMARY:
This study is a single-center, open, dose-escalation Phase I clinical study. It is designed to evaluate the safety, tolerability, preliminary efficacy and immunogenicity of treating NV-001, a king of hybrid-membrane-based tumor vaccine in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a single-center, open, dose-escalation Phase I clinical study. It is designed to evaluate the safety, tolerability, preliminary efficacy and immunogenicity of treating NV-001, a king of hybrid-membrane-based tumor vaccine in patients with advanced solid tumors. The patients will be treated with vaccines generated based on their tumor tissues.Various doses will be tested according to the protocol to get preliminary safety and efficacy evidence.

ELIGIBILITY:
Inclusion Criteria:

* patients with histopathologically and/or cytologically confirmed non-surgically resectable advanced/metastatic solid tumors.
* patients with progression on prior standard treatment regimens or intolerance to standard treatment or no standard treatment.
* an Eastern Cooperative Oncology Group (ECOG) Physical Status (PS) score of 0 or 1 and an expected survival time of ≥12 weeks
* confirmed clinical or imaging progression after the most recent antitumor therapy: at least 1 measurable lesion according to RECIST 1.1 criteria.
* Substantially normal major organ function and screening laboratory values that meet the following criteria:

A. Bone marrow function: absolute neutrophil count ≥ 1000/μL; hemoglobin ≥ 9g/dL; platelet count ≥ 75,000/μL.

B. Liver function: serum total bilirubin ≤ 1.5 x upper limit of normal (ULN); serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 x ULN (patients with liver metastases should be ≤ 5 x ULN); alkaline phosphatase < 2.5 x ULN (patients with liver and bone involvement should be ≤ 5 x ULN).

C. Renal Function: Serum creatinine ≤ 2.5 x ULN, or creatinine clearance ≥ 30 mL/min, whether actually measured by urine collection or estimated using the Cockcroft-Gault formula.

D. coagulation: prothrombin time (PT), International Normalized Ratio (INR), and Partial Thromboplastin Time (PTT) ≤ 1.5 × ULN.

* presence of biopsy lesions with acceptable clinical risk or lesions amenable to palliative surgical resection. Presence of a tumor lesion amenable to tumor tissue biopsy.
* have an expected survival of more than 12 weeks.
* the patient understands and complies with the study protocol and has signed the appropriate Informed Consent Form (ICF), which must be signed prior to the study procedure. 11. for patients of childbearing potential, the patient must be able to understand and comply with the study protocol.
* For patients of childbearing potential: Patients should agree to use effective contraception during treatment and for at least 90 days after the last dose of study treatment, including double-barrier contraception, condoms, contraceptive pills or injectables, and intrauterine devices (IUDs). Male patients should agree to avoid sperm donation.

Exclusion Criteria:

* has received other systemic antitumor therapy within 28 days or 5 half-lives prior to the first treatment. or has not recovered from the previous treatment (all three cases, whichever is longer);
* has received radiotherapy within 14 days prior to the first dose.
* has received a live or live attenuated vaccine within 30 days prior to the first dose.
* use of immunosuppressive drugs currently or within 14 days prior to the first dose.
* has had major surgery within 28 days or non-study related minor surgery within 7 days prior to the first dose.
* the patient has a history of allergic or hypersensitivity reactions to any of the components of NV-001.
* female patients who are breastfeeding or have a positive serum pregnancy test at the time of the screening visit.
* insufficient biopsy to complete the experiment
* any Grade 4 immune-related AE (irAE) on prior immunotherapy (patients with endocrine disorders receiving replacement therapy or experiencing asymptomatic elevations in serum amylase or lipase are eligible for enrollment), any irAE on prior immunotherapy that resulted in permanent discontinuation of therapy, or any Grade 3 irAE within ≤ 6 months prior to initiation of treatment.
* prior toxicity from antineoplastic therapy that remains at NCI-CTCAE ≥ Grade 2 (except for alopecia, vitiligo, and experimental indications of Grade 2 or higher as defined in the Inclusion Criteria); subjects with neurotoxicity ≥ Grade 2 may be eligible for enrollment at the discretion of the Investigator; subjects with irreversible toxicity may be eligible for enrollment at the discretion of the Investigator.
* the presence of clinically significant pulmonary fibrosis or interstitial pneumonitis as determined by the investigator.
* the presence of clinically significant severe ophthalmic disease as determined by the investigator based on screening ophthalmologic examination.
* the presence of other malignant tumors within the previous 5 years, with the exception of cured basal cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the breast, and carcinoma in situ of the cervix.

prolonged use (≥14 consecutive days) of immunosuppressive or other immunomodulatory drugs (e.g., corticosteroids: prednisone or equivalent) within 6 months, except that topical medications (e.g., ointments, eye drops, inhalers, or nasal sprays) are permitted, and topical medications must not exceed the dose recommended in the insert or if there are any signs of systemic exposure; or other acquired or congenital immunodeficiency diseases; or History of organ transplantation.

* the presence of clinically symptomatic central nervous system tumors or metastases.
* the presence of an active infection including tuberculosis (documented history, investigator judgment and radiology, and local laboratory testing), hepatitis B (hepatitis B surface antigen positive, HBV DNA above the lower limit of detection), hepatitis C (HCV antibody positive, HCV RNA positive), HIV (HIV antibody positive), and enrolled patients with viral load-negative HBV or HCV who have consented to Antiviral therapy and/or regular viral indicator monitoring as determined by the physician.
* documented primary immunodeficiency or organ transplantation.
* subjects with a history of active gastrointestinal bleeding, hemoptysis or hemorrhage.
* other conditions that may result in increased risk associated with the study medication, or affect compliance with the trial, which in the opinion of the investigator make participation in this trial inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing dose-limiting toxicities (DLTs) | in the first 28 days after the first dose.
  Number of Participants Experiencing dose-limiting toxicities (DLTs)
Number of Participants Experiencing Adverse Events (AEs) | From signed ICF until the date of last visit or start new antitumor therapy, whichever comes first, assessed up to 36 months
  Number of Participants Experiencing Adverse Events (AEs)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 36 month
  Overall Response Rate (ORR)
Disease Control Rate(DCR) | Up to 36 month
  Disease Control Rate(DCR)

OTHER OUTCOMES:
Progression-Free Survival (PFS) | Up to 36 month
  Progression-Free Survival (PFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No